CLINICAL TRIAL: NCT02793310
Title: Corneal Transplantation by DMEK - is it Really Better Than DSAEK?
Brief Title: DMEK Versus DSAEK Study
Acronym: DMEK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL55972.068.15
Record Dates: First submitted 2016-05-20; First posted 2016-06-08 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Fuchs' Endothelial Dystrophy
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DMEK (Active Comparator): The intervention group will receive cornea transplantation by DMEK
  Interventions: Procedure: DMEK
- DSAEK (Active Comparator): The usual care / control group will receive cornea transplantation by DSAEK
  Interventions: Procedure: DSAEK

INTERVENTIONS:
Procedure: DMEK — The intervention group will receive cornea transplantation by DMEK
  Arms: DMEK
Procedure: DSAEK — The usual care / control group will receive cornea transplantation by DSAEK
  Arms: DSAEK

SUMMARY:
The purpose of this study is to determine whether corneal transplantation by Descemet Membrane Endothelial Keratoplasty more favourable and cost-effective is compared to Descemet Stripping Automated Endothelial Keratoplasty for Fuchs Endothelium Corneal Dystrophy.

DETAILED DESCRIPTION:
FECD is a progressive, multifactorial and irreversible disease characterized by accelerated loss of corneal endothelial cells in the innermost layer of the cornea that leads to vision impairment and potential blindness if left untreated. FECD is responsible for more than 50% of the 1.300 annual corneal transplantations in the Netherlands.

Corneal transplantation improves vision and quality of life in patients with corneal disease. Currently, the standard of care for patients with Fuchs Endothelial Corneal Dystrophy (FECD) is Descemet Stripping Automated Endothelial Keratoplasty (DSAEK), in which only the posterior layers of the cornea are transplanted. However, visual recovery following DSAEK is suboptimal. Descemet Membrane Endothelial Keratoplasty (DMEK), the latest technique in corneal transplantation involves transplantation of only a monolayer of corneal endothelium and Descemet's membrane providing the thinnest endothelial graft possible. DMEK has been suggested to result in faster and better visual recovery compared to DSAEK. While the economic burden, both medical and social, from this disease has not been assessed to date, costs associated with corneal transplantation reach $ 110 million dollars yearly for the 47.000 transplantations in the USA.

The objective of this project is to assess the effects and costs of DMEK vs. DSAEK in order to determine whether the new technique is effective and cost-effective over the standard technique.

The primary outcome measure is best-corrected visual acuity. Secondary outcome measures are contrast acuity, astigmatism, quality of vision, endothelial cell loss, incidence of graft rejection, primary graft failure, cornea donor loss due to preparation, and generic and vision-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Cornea decompensation caused Fuchs Endothelial Corneal Dystrophy

Exclusion Criteria:

* Ocular comorbidities other than cataract
* Previous corneal transplantation
* Human leukocyte antigen (HLA) matched keratoplasty
* Inability to complete follow-up

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Change in best-corrected visual acuity | Preoperatively and 3, 6, 12 months post-operatively
  Visual acuity will be measured by ETDRS letter charts

SECONDARY OUTCOMES:
Change in contrast sensitivity | Preoperatively and 3, 6, 12 months post-operatively
  Contrast sensitivity will be measured using the CSV-1000 chart by Vector Vision
Change in astigmatism | Preoperatively and 3, 6, 12 months post-operatively
  Astigmatism will be measured using the The Pentacam HR (Oculus Inc., Lynnwood, USA)
Change in corneal scatter | Preoperatively and 3, 6, 12 months post-operatively
  Corneal scatter will be measured using a confocal microscope
Change in endothelial cell loss | Preoperatively and 3, 6, 12 months post-operatively
  Endothelial cell loss will be measured using specular microscopy photography.
Incidence of graft rejection | 3, 6, 12 months post-operatively
Incidence of primary graft failure | 3, 6, 12 months post-operatively
  Primary Graft failure will be assessed during ophthalmic examination.
Incidence of cornea donor loss due to preparation | Preoperatively
  The eye bank providing the donor cornea's will register cornea donor loss if a complication occurs during preparation that renders the cornea unusable.
Change in generic quality of life | Preoperatively and 3, 6, 12 months post-operatively
  Generic quality of life will be measured using the HUI3 (Health Utility Index Mark 3), which test 8 dimensions: vision, hearing, speech, ambulation, dexterity, emotion, cognition and pain.
Change in generic quality of life | Preoperatively and 3, 6, 12 months post-operatively
  Generic quality of life will be measured using the EQ-5D-5L questionnaire, which tests 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
Change in vision-related quality of life | Preoperatively and 3, 6, 12 months post-operatively
  Vision-related quality of life will be measured using the National Eye Institute Visual Function Questionnaire (NEI VFQ-25), which is specified for vision-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Rudy Nuijts, PhD, Principal Investigator — Department of Ophthalmology, Maastricht University Medical Centre
Locations (1):
- Maastricht University Medical Centre, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gipson IK. Age-related changes and diseases of the ocular surface and cornea. Invest Ophthalmol Vis Sci. 2013 Dec 13;54(14):ORSF48-53. doi: 10.1167/iovs.13-12840. PMID 24335068
- See also: Nederlandse Orgaan Transplantatie Register (NOTR) — http://www.transplantatiestichting.nl/